CLINICAL TRIAL: NCT05477563
Title: A Phase 3b Study to Evaluate Efficacy and Safety of a Single Dose of Autologous CRISPR Cas9 Modified CD34+ Human Hematopoietic Stem and Progenitor Cells (CTX001) in Subjects With Transfusion-Dependent β-Thalassemia or Severe Sickle Cell Disease
Brief Title: Evaluation of Efficacy and Safety of a Single Dose of CTX001 in Participants With Transfusion-Dependent β-Thalassemia and Severe Sickle Cell Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX21-CTX001-161; 2024-514641-12-00 (Other: EU CT number)
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-03

CONDITIONS: Beta-Thalassemia; Thalassemia; Hematologic Diseases; Genetic Diseases, Inborn; Hemoglobinopathies; Sickle Cell Disease; Sickle Cell Anemia
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Hematologic Diseases; Genetic Diseases, Inborn; Hemoglobinopathies; Anemia, Sickle Cell | interventions — exagamglogene autotemcel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX001 (Experimental): CTX001 (autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the erythroid lineage-specific enhancer of the BCL11A gene). Participants will receive a single infusion of CTX001 through a central venous catheter.
  Interventions: Biological: CTX001

INTERVENTIONS:
Biological: CTX001 — Administered by intravenous (IV) infusion following myeloablative conditioning with busulfan
  Other Names: Exagamglogene autotemcel; Exa-cel

SUMMARY:
This is a single-dose, open-label study in participants with transfusion-dependent β-thalassemia (TDT) or severe sickle cell disease (SCD). The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 modified CD34+ human hematopoietic stem and progenitor cells (hHSPCs) using CTX001.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with TDT and SCD:
* Eligible for autologous stem cell transplant as per investigator's judgment.
* Participants with TDT:
* Diagnosis of TDT as defined by:
* Documented homozygous β-thalassemia or compound heterozygous β-thalassemia including β-thalassemia/hemoglobin E (HbE). Participants can be enrolled based on historical data, but a confirmation of the genotype using the study central laboratory will be required before busulfan conditioning
* History of at least 100 milliliter (mL)/kilograms (kg)/year or 10 units/year of packed red blood cells (RBC) transfusions in the prior 2 years before signing the consent or the last rescreening for patients going through re-screening
* Participants with SCD:
* Diagnosis of severe SCD as defined by:
* Documented SCD genotypes
* History of at least two severe VOCs events per year for the previous two years prior to enrollment

Key Exclusion Criteria:

* Participants with TDT and SCD:
* A willing and healthy 10/10 human leukocyte antigen (HLA)-matched related donor is available per investigator's judgement
* Prior hematopoietic stem cell transplant (HSCT)
* Clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by the investigator
* Participants with TDT:
* Participants with associated α-thalassemia and >1 alpha deletion, or alpha multiplications
* Participants with sickle cell β-thalassemia variant
* Participants with SCD:
* History of untreated moyamoya syndrome or presence of moyamoya syndrome at screening

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2027-06-09 (Estimated); Study Completion 2027-06-09 (Estimated)

PRIMARY OUTCOMES:
Fetal Hemoglobin (HbF) Concentration Over Time | Up to 12 Months After CTX001 Infusion
Total Hemoglobin (Hb) Concentration Over Time | Up to 12 Months After CTX001 Infusion

SECONDARY OUTCOMES:
TDT and SCD: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Signing of Informed Consent up to 12 Months After CTX001 Infusion
TDT and SCD: Proportion of Participants With Engraftment (First day of 3 Consecutive Measurements of Absolute Neutrophil Count (ANC) >=500 per Microliter [mcgL] on 3 Different Days) | Within 42 Days After CTX001 Infusion
TDT and SCD: Time to Engraftment | Up to 12 Months After CTX001 Infusion
TDT and SCD: Incidence of Transplant-Related Mortality (TRM) Within 100 Days After CTX001 Infusion | Within 100 Days After CTX001 Infusion
TDT and SCD: Incidence of TRM Within 12 Months After CTX001 Infusion | Within 12 Months After CTX001 Infusion
TDT and SCD: Incidence of All-cause Mortality | From Signing of Informed Consent up to 12 Months After CTX001 Infusion
TDT and SCD: Relative Reduction in Annualized Volume of RBC Transfusions | From Day 60 up to 12 Months After CTX001 Infusion
TDT and SCD: Proportion of Alleles With Intended Genetic Modification Present in Peripheral Blood Over Time | Up to 12 Months After CTX001 Infusion
TDT and SCD: Proportion of Alleles With Intended Genetic Modification Present in CD34+ Cells of the Bone Marrow Over Time | Up to 12 Months After CTX001 Infusion
TDT: Duration Transfusion Free in Participants | Up to 12 Months After CTX001 Infusion
SCD: Relative Reduction in Annualized Rate of Severe Vaso-Occlusive Crises (VOCs) | From Baseline up to 12 Months After CTX001 Infusion
SCD: Relative Reduction in Annualized Rate of Inpatient Hospitalizations for Severe VOCs | From Baseline up to 12 Months After CTX001 Infusion
SCD: Relative Reduction in Annualized Duration of Hospitalization for Severe VOCs | From Baseline up to 12 Months After CTX001 Infusion
SCD: Relative Reduction in Haptoglobin | From Baseline up to 12 Months After CTX001 Infusion
SCD: Relative Reduction in Lactate dehydrogenase | From Baseline up to 12 Months After CTX001 Infusion
SCD: Relative Reduction in Total Bilirubin | From Baseline up to 12 Months After CTX001 Infusion
SCD: Relative Reduction in Indirect Bilirubin | From Baseline up to 12 Months After CTX001 Infusion

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - New York Presbyterian Hospital - Morgan Stanley Children's Hospital, New York, New York
  - Levine Children's Hospital - Hematology, Charlotte, North Carolina
  - TriStar Medical Group Children's Specialists - Pediatric Oncology, Nashville, Tennessee
- University Hospital Dusseldorf - Department of Pediatric Oncology, Hematology and Clinical Immunology, Düsseldorf, Germany
- IRCSS Ospedale Pediatrico Bambino Gesu - Dipartimento di Onco-Ematologia e Terapia Cellulare e Genica, Rome, Italy
- King Faisal Specialist Hospital & Research Centre - Riyadh - Hematology, Al Mathar Ash Shamali, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/